CLINICAL TRIAL: NCT00206830
Title: SHORTness of Breath In the Emergency Department (SHORTIE)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abbott RDx Cardiometabolic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 011
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Acute Myocardial Infarction; Heart Failure; Pulmonary Embolism
MeSH Terms: conditions — Heart Failure; Pulmonary Embolism

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Control-Blinded from Results (No Intervention)
- Access to Results (Experimental)
  Interventions: Device: Triage Profiler S.O.B. Panel

INTERVENTIONS:
Device: Triage Profiler S.O.B. Panel
  Arms: Access to Results

SUMMARY:
SHORTIE is a two-phase study to determine the impact of the Triage Profiler S.O.B. (Shortness Of Breath) Panel on patient management, outcome, and cost.

DETAILED DESCRIPTION:
Patients presenting to the ED with a primary complaint of shortness of breath will a have blood sample collected at enrollment and tested using the Triage® Profiler S.O.B. Panel (measuring creatine kinase MB [CK-MB], myoglobin, troponin I, B-type natriuretic peptide [BNP], D-dimer). The test is used as an aid in the diagnosis of myocardial infarction (MI), an aid in the diagnosis and assessment of severity of heart failure (HF), and an aid in the assessment and evaluation of disseminated intravascular coagulation including pulmonary embolism (PE). Phase I is an observational study and results of the Triage Profiler S.O.B. panel will be blinded to all attending physicians and health care workers. In Phase II, patients will be assigned to either the experimental arm or the control arm of the study. In the experimental arm, the Triage Profiler S.O.B. Panel results will be available to the treating physician and can be incorporated into the decision making process. In the control arm, treating physicians and staff will be blinded to the Triage Profiler S.O.B. Panel results. Time to appropriate treatment, length of ED stay, patient outcome and hospital costs will be assessed in all patients and used to determine the impact of Triage Profiler S.O.B Panel on these parameters. Furthermore, the diagnostic accuracy of the Triage Profiler S.O.B Panel will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older.
* Visit to the ED is due to a primary complaint of shortness of breath alone or shortness of breath with associated chest pain, cough or edema.

Exclusion Criteria:

* Blood sample cannot be collected before treatment is initiated, specifically CPR or treatment with i.v. diuretics, injectable anticoagulants, thrombolytics
* Patient is unwilling or unable to give consent to participate in the study
* Patient has renal disease requiring dialysis
* Patients with a clear exacerbation of isolated asthma
* Patients with trauma that interferes with normal breathing function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306
Dates: Start 2005-04; Primary Completion 2006-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Time to specific treatment for final diagnosis
Length of stay in the emergency department (ED)
ED and total hospital costs

SECONDARY OUTCOMES:
Outcome at 30 days (Phase I and II) and 90 days (Phase II)
Diagnostic accuracy of the Triage® Profiler S.O.B. panel for acute myocardial infarction (AMI), heart failure (HF) and pulmonary embolism (PE) in patients presenting with S.O.B.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Maisel, MD, Principal Investigator — VA, University of California, San Diego
Locations (5):
- United States (5):
  - University of Massachusetts Medical Center USA, Worcester, Massachusetts
  - New York Methodist Hospital, Brooklyn, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Duke University Hospital Durham, Durham, North Carolina
  - Hospital of the Univ. of Pennsylvania, Philadelphia, Pennsylvania